CLINICAL TRIAL: NCT04294004
Title: A Prospective, Randomized and Non-randomized, Controlled, Single-blind and Open-label, Dose-finding, Multi-center, Parallel Group Study of Safety/Efficacy of KUR-113 Bone Graft Versus Local Autograft for the Treatment of Single-level Transforaminal Lumbar Interbody Fusion
Brief Title: KUR-113 Bone Graft Versus Local Autograft for the Treatment of Single-level Transforaminal Lumbar Interbody Fusion
Acronym: STRUCTURE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Avania (Industry); Kuros BioSciences B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUR-113/01
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Degenerative Disc Disease; Spinal Fusion
Keywords: Spinal Fusion; Posterolateral Fusion; MagnetOs; Fibrin-PTH (KUR-113)
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Fibrin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Due to the different technical procedures between the control and the intervention arms (KUR-113 Bone Graft versus local autograft), investigators cannot be blinded to the treatment. However, all stage 1 patients will remain blinded for the duration of their participation in the study. All stage 2 patients will receive the same treatment and will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KUR-113, Stage 1 (Experimental): During stage 1, subjects randomized to this arm will receive TGplPTH1-34 in fibrin (0.4mg/ml) that will be applied within and around a polyetheretherketone (PEEK) intervertebral cage. The maximum dose that will be applied is 4 mg of TGplPTH1-34 in 10mL KUR-113 Bone Graft.
  Interventions: Combination Product: TGplPTH1-34 in fibrin
- Autologous Bone Graft (Active Comparator): During stage 1 of the study, subjects randomized to this arm will receive local autologous bone graft. In the event of insufficient local autograft, Iliac crest bone graft may be used to supplement.
  Interventions: Other: Autologous Bone Graft
- KUR-113, Stage 2 (Experimental): During stage 2, subjects will receive TGplPTH1-34 in fibrin that will be applied within and around a PEEK intervertebral cage at a concentration of 0.7mg/ml. The concentration received was selected by the DSMB based on the results of stage 1. The maximum dose that will be applied is 7 mg of TGplPTH1-34 in 10mL KUR-113 Bone Graft.
  Interventions: Combination Product: TGplPTH1-34 in fibrin

INTERVENTIONS:
Combination Product: TGplPTH1-34 in fibrin — TGplPTH1-34 within a fibrin matrix applied within and around a polyetheretherketone (PEEK) intervertebral cage
  Other Names: KUR-113
  Arms: KUR-113, Stage 1; KUR-113, Stage 2
Other: Autologous Bone Graft — Local autograft collected from decompression which may be supplemented with iliac crest bone graft (ICBG) if local autograft is insufficient.
  Arms: Autologous Bone Graft

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of KUR-113 Bone Graft (TGplPTH1-34 in fibrin) compared to local autograft for the treatment of Degenerative Disk Disease (DDD).

DETAILED DESCRIPTION:
Degenerative disc disease (DDD) is a common disorder of the lumbar spine. Clinically, DDD causes discogenic back pain and may cause related radicular, neuropathic, claudicatory, and referred pain.

This is a prospective, randomized and non-randomized, controlled, single-blind and open-label, dose-finding, multi-center study which intends to demonstrate the safety and efficacy of KUR-113 Bone Graft (TGplPTH1-34 in fibrin) versus local autograft. The study will enroll 50 patients with Degenerative Disk Disease (DDD) requiring single-level interbody fusion along with posterolateral fusion (PLF) with posterior fixation who meet eligibility criteria and agree to participate in the study. Safety and efficacy of KUR-113 Bone Graft will be evaluated by analyzing all clinical as well as radiological endpoints and adverse events. This phase 2a study is not powered to detect non-inferiority. All patients will undergo clinical and radiological assessments at initial hospital discharge (on average 3 days post-surgery), 6 weeks, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by the patient.
2. Male or female patient ≥ 25 up to and including 75 years old. Females of childbearing potential with a negative urine pregnancy test at Screening. Females of childbearing potential must agree to use acceptable contraception for at least 12 months after surgery and investigational product placement.
3. Patients with degenerative disc disease with up to grade 1 spondylolisthesis and with leg pain requiring up to 3 levels of laminectomy/decompression and a single-level fusion (L2 - S1). DDD is defined by the presence of one or more of the following:

   1. instability (angulation ≥ 5 degrees or translation ≥ 3 mm on flexion/extension radiographs),
   2. osteophyte formation of facet joints or vertebral endplates,
   3. decreased disc height by > 2 mm, but dependent upon the spinal level,
   4. scarring/thickening of ligamentum flavum, annulus fibrosis or facet joint capsule,
   5. disc degeneration and/or herniation,
   6. facet degeneration,
   7. vacuum phenomenon.
4. Patients with an Oswestry Disability Index (ODI) score ≥ 35.
5. Patients with a Visual Analogue Scale (VAS) leg score ≥ 40.
6. Failed conservative treatment (physical therapy, bed rest, medications, spinal injections or transcutaneous electrical nerve stimulation) for a period of 6 months prior to study enrollment.
7. Patients willing to undergo PK sampling.

Exclusion Criteria:

1. Patients with open epiphyseal plates.
2. Patient requiring emergency spinal decompression or spinal fusion.
3. Patients requiring multilevel fusion or expected to need secondary intervention within one year following surgery.
4. Any prior fusion or attempted fusion at an adjacent level.
5. Any prior fusion or attempted fusion at the index level.
6. Pregnant or breast-feeding women.
7. Known or suspected allergies to any of the components of KUR-113 Bone Graft (e.g.

   hypersensitivity to aprotinin).
8. Any prior use of teriparatide or abaloparatide or graft material containing PTH1-34.
9. Patients with hypercalcemic disorders (e.g., primary hyperparathyroidism).
10. Patients with Paget's Disease or unexplained high levels of alkaline phosphatase.
11. Prior radiation therapy involving bone.
12. Medical history or radiographic evidence of a metabolic bone disorder (e.g. Paget's Disease) or other condition that would negatively impact the healing process.
13. Any medical condition requiring radiotherapy or immunosuppression.
14. History of thyroid autoimmune disease (Hashimoto's thyroiditis, Graves' disease) or hyperthyroidism.
15. Patients on chronic systemic steroids (i.e. > 14 consecutive days) within 6 months prior to Screening Visit.
16. Osteopenia (T score < -1.0) or osteoporosis of the spine (T score < -2.5).
17. DDD related to benign or malignant tumor.
18. History or presence of active malignancy.
19. Hereditary disorders predisposing to osteosarcoma.
20. Patients with invasive skin cancer.
21. Evidence of local or systemic infection.
22. Patients with known active COVID-19 disease.
23. Current smokers.
24. Type 1 diabetes (regardless of HbA1c) or Type 2 diabetes with a documented HbA1c > 7.0.
25. Any acute or chronic concurrent medical conditions that in the Investigator's opinion are a contraindication to the procedure and study participation.
26. Participation in another investigational study within 30 days prior to surgery for investigational devices, or within the last three months for investigational drugs. (Note: trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).
27. Known substance abuse, psychiatric disorder or a condition which, in the opinion of the investigator, may influence the healing or ability to comply with protocol requirements.
28. Involved in active litigation relating to his/her spinal condition or workers compensation claimants.
29. BMI greater than 40.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic interbody fusion | Month 12 post-surgery
  Evidence of bridging trabeculae or continuous bony connection between superior and inferior vertebral body on CT-scan as determined by an independent radiology expert panel (IREP).

SECONDARY OUTCOMES:
Composite Endpoint | Month 6 and Month 12 post-surgery
  Radiographic interbody fusion using CT-scans, functional outcome (decrease of 15 points or more on Oswestry Disability Index (ODI)) and no post-surgical intervention to aid fusion or replace any of the spinal implants.
Radiographic interbody fusion | Month 6 post-surgery
  Determined by IREP using CT-scans
Radiographic posterolateral fusion | Month 6 and Month 12 post-surgery
  Determined by IREP using CT-scans
ODI | Week 6, Month 3, Month 6, Month 12, and Month 24 post-surgery
  Change from baseline
Leg Pain | Initial discharge from hospital (on average 3 days post-surgery), Week 6, Month 3, Month 6, Month 12, and Month 24 post-surgery
  Change from baseline using Visual Analogue Scale (VAS). VAS is scored from 0 to 100 with higher numbers being a worse outcome than a lower number.
Back Pain | Initial discharge from hospital (on average 3 days post-surgery), Week 6, Month 3, Month 6, Month 12, and Month 24 post-surgery
  Change from baseline using Visual Analogue Scale (VAS). VAS is scored from 0 to 100 with higher numbers being a worse outcome than a lower number.
Number of Secondary Interventions | Up to Month 24 post-surgery
  Revisions, re-operations, removals, supplemental fixations, or any other procedure that adjusts or in any way removes part of the original implant configuration with or without replacement of the components

CONTACTS AND LOCATIONS:
Overall Officials: John Chi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (15):
- United States (15):
  - University of California San Diego, La Jolla, California
  - Justin Parker Neurological Institute, Boulder, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University-Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Kansas Spine and Specialty Hospital, Wichita, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Orthopedic Associates of Michigan, Grand Rapids, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - University at Buffalo Neurosurgery, Williamsville, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - South Texas Spine Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No